CLINICAL TRIAL: NCT00789087
Title: Analysis of Clinical and Radiological Results of Two Methods of Talc Pleurodesis in Patients With Recurrent Malignant Pleural Effusion
Brief Title: Talc Pleurodesis in Patients With Recurrent Malignant Pleural Effusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Ricardo M. Terra, University of São Paulo Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1105/04
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2008-11-11 (Estimated); Status verified 2008-11

CONDITIONS: Recurrent Malignant Pleural Effusion.
Keywords: Pleural Effusion.; Talc.; Pleurodesis.; Quality of Life.; Thoracoscopy.
MeSH Terms: conditions — Pleural Effusion, Malignant; Pleural Effusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Videothoracoscopic talc poudrage (VT) (Active Comparator)
  Interventions: Procedure: Videothoracoscopic talc poudrage (VT).
- 2. Talc slurry through a chest tube (DT) (Active Comparator)
  Interventions: Procedure: Talc slurry through a chest tube (DT).

INTERVENTIONS:
Procedure: Videothoracoscopic talc poudrage (VT). — Videothoracoscopic talc poudrage
  Other Names: Videothoracoscopic talc poudrage
  Arms: 1. Videothoracoscopic talc poudrage (VT)
Procedure: Talc slurry through a chest tube (DT). — Talc slurry through a chest tube
  Other Names: Talc slurry through a chest tube
  Arms: 2. Talc slurry through a chest tube (DT)

SUMMARY:
The purpose of this study is to analyze and compare radiological lung expansion after talc pleurodesis performed either by videothoracoscopy or chest tube and correlate it with clinical outcome. Secondary endpoints evaluated were: clinical efficacy, safety, quality of life and survival.

DETAILED DESCRIPTION:
Talc pleurodesis is the most popular method to control symptoms of recurrent malignant pleural effusion. The intrapleural talc delivery may be by videothoracoscopy and talc poudrage or talc slurry thought a chest tube and the best method is still controversial. Although the lung expansion is a key criteria for success of the procedure, its characteristics are poorly studied.

Patients were enrolled into two groups: videothoracoscopic talc poudrage (VT) and talc slurry through a chest tube (DT). Lung expansion was evaluated through chest CT scans obtained obtained in the first 7 days and 1, 3 and 6 months after pleurodesis. All examinations were revised by two independent observers. Clinical efficacy (considered as lack of new procedures during follow up), complications, drainage duration, hospital stay and quality of life (general and specific questionnaires) were also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Malignant pleural effusion confirmed by cytological analysis of pleural fluid and/or pleural biopsy;
* Recurrent pleural effusion with symptoms;
* Chest radiography with lung expansion after thoracocentesis;
* Karnofsky Performance Status > 70;
* Written informed patient consent were obtained.

Exclusion Criteria:

* Hemorrhagic diathesis;
* Active infection;
* Cutaneous infiltration;
* Patients unable to understand the questionnaires;
* Age: > 90 yo or < 18 yo.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Radiological lung expansion after talc pleurodesis and clinical outcome | 6 months

SECONDARY OUTCOMES:
Clinical efficacy, safety, quality of life and survival. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo M. Terra, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Terra RM, Junqueira JJM, Teixeira LR, Vargas FS, Pego-Fernandes PM, Jatene FB. Is full postpleurodesis lung expansion a determinant of a successful outcome after talc pleurodesis? Chest. 2009 Aug;136(2):361-368. doi: 10.1378/chest.08-2448. Epub 2009 Apr 6. PMID 19349389